CLINICAL TRIAL: NCT06704256
Title: SCM Muscle as a Marker for Frailty in Patients Undergoing ENT Surgery
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Mingyang L Gray, Assistant Professor Facial Plastic and Reconstructive Surgery Department of Otolaryngology - Head and Neck Surgery, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-24-00751
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients Undergoing Non-Oncologic and Neck surgery: Non-oncologic patients presenting for head and neck surgery with available neck CT scans.

SUMMARY:
This study focuses on evaluating the relationship between physical frailty and measurements of the muscles of the neck in patients undergoing non-cancer Head and Neck surgery.

ELIGIBILITY:
Inclusion Criteria:

• Non-oncologic patients presenting for head and neck surgery with available neck CT scans.

Exclusion Criteria:

* Patients undergoing cancer surgery
* Patients under18 years of age
* Patients without pre-surgical CT-scans of the head and neck

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Non-oncologic patients presenting for head and neck surgery with available neck CT scans
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2026-10-23 (Estimated); Study Completion 2026-10-23 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle size | End of study at 6 months
  Skeletal muscle derived measures of size of neck skeletal musculature. No maximum or minimum.
Skeletal muscle density | End of study at 6 months
  Skeletal muscle derived measures of density of neck skeletal musculature. No maximum or minimum.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Hernandez, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  Any purpose. Data are available indefinitely at (Link to be included in the URL field below).